CLINICAL TRIAL: NCT07274826
Title: Intact Potential Symptoms and Biomarker Analysis in Diagnosis of Acid Sphingomyelinase Deficiency (ASMD)
Brief Title: Diagnostic Creteria of Acid Sphingomyelinase Deficiency (ASMD)
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Nasser Aly, MD, Sohag University
Other Study IDs: Soh_Med_25_9____17MS
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Acid Sphingomyelinase Deficiency (ASMD)
Keywords: ASMD; Neiman _PICK disease
MeSH Terms: conditions — Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acid sphingomyelinase Deficiency known as Neiman _PICK disease is a group of rare genetic diseases. This study includes analysis of clinical manifestations in patients with ASMD and investigations done for diagnosis of these patients

ELIGIBILITY:
Inclusion Criteria:

* all patients diagnosed with ASMD in Sohag

Exclusion Criteria:

* Patients with hepatosplenomegaly due to other cause Patients who refuse consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients diagnosed with Niemann _PICK disease specifically confirmed through clinical evaluation, biochemical testing and genetic analysis, receiving follow up and clinical care at hematology and git and metabolic centre's in Sohag Patients may present with variable neurological, visceral, or systemic manifestations characteristic of Niemann _PICK disease.
  Recruitment will include both newly diagnosed and previously diagnosed who meet the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-08-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
spleen volumes measured by US expressed relative to basaline for each patient | From basaline to month 12
  Change in spleen volumes following treatment over 12months study period

SECONDARY OUTCOMES:
Liver size measured by ultrasound | Basaline, weak 12,weak 24
  Changes in liver volume

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No